CLINICAL TRIAL: NCT07054515
Title: 18-month Double-blind, Randomized, Placebo-controlled, Multicenter, Phase 3 Study to Evaluate the Safety and Efficacy of Oral Nizubaglustat (AZ-3102) in Late-infantile and Juvenile Forms of Niemann-Pick Type C Disease and in Late-infantile and Juvenile-onset Forms of GM1 Gangliosidosis or GM2 Gangliosidosis
Brief Title: A Study to Evaluate the Safety and Efficacy of Oral Nizubaglustat (AZ-3102) in Late-infantile and Juvenile Forms of Niemann-Pick Type C Disease, GM1 Gangliosidosis or GM2 Gangliosidosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Azafaros A.G. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZA-001-301; 2024-515778-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-09

CONDITIONS: Niemann-Pick Type C Disease; GM1 Gangliosidosis; GM2 Gangliosidosis
Keywords: Nizubaglustat
MeSH Terms: conditions — Niemann-Pick Disease, Type C; Gangliosidosis, GM1; Gangliosidoses, GM2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, other study personnel at the site, and the Sponsor will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subprotocol NCT07082725: Intervention Group NPC (Experimental): Participants will be randomized to receive either nizubaglustat or placebo at a 2:1 ratio (nizubaglustat:placebo)
  Interventions: Drug: AZ-3102; Drug: Placebo
- Subprotocol NCT07082543: Intervention Group GM1/GM2 (Experimental): Participants will be randomized to receive either nizubaglustat or placebo at a 2:1 ratio (nizubaglustat:placebo)
  Interventions: Drug: AZ-3102; Drug: Placebo

INTERVENTIONS:
Drug: AZ-3102 — Oral dispersible tablets
  Other Names: nizubaglustat
Drug: Placebo — A matching placebo will be administered in the same regimen as the intervention

SUMMARY:
An 18-month double-blind, randomized, placebo-controlled, multicenter, Phase 3 study to evaluate the safety and efficacy of oral nizubaglustat (AZ-3102) in late-infantile and juvenile forms of Niemann-Pick type C disease and in late-infantile and juvenile-onset forms of GM1 gangliosidosis or GM2 gangliosidosis

DETAILED DESCRIPTION:
This is a Phase 3 randomized, double-blinded, placebo-controlled study that will evaluate the safety and efficacy of oral nizubaglustat (AZ-3102) in multiple disease areas using a Master Protocol Research Program. Participants are randomized to different subprotocols based on disease type: Niemann-Pick type C (NPC), GM1 gangliosidosis or GM2 gangliosidosis.

Treatment specific procedures will be described in the disease-specific subprotocol. Individual subprotocols may have additional eligibility requirements, safety and efficacy procedures, or endpoints, which will be described in the corresponding subprotocols.

For information specific to each individual subprotocol included in this trial, please refer to the corresponding, separate, clinicaltrials.gov records: Niemann-Pick type C disease NCT07082725 and GM1 gangliosidosis or GM2 gangliosidosis NCT07082543.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants, aged 4 years and older with a diagnosis of the late-infantile or juvenile form of NPC disease. Detailed inclusion criteria are presented in the NPC disease-specific subprotocol AZA-001-301-NPC (NCT07082725).
* Male and female participants, aged 4 years and older with a diagnosis of GM1 or GM2 (Tay-Sachs, Sandhoff, or GM2AB variant disease) gangliosidosis of late-infantile/ juvenile onset. Detailed inclusion criteria are presented in the GM1/GM2 gangliosidosis-specific subprotocol AZA-001-301-GMx (NCT07082543).

Exclusion Criteria:

* Detailed exclusion criteria are presented in the NPC disease-specific subprotocol AZA-001-301-NPC
* Detailed exclusion criteria are presented in the GM1/GM2 gangliosidosis-specific subprotocol AZA-001-301-GMx

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2027-11-04 (Estimated); Study Completion 2027-11-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants allocated to subprotocol AZA-001-301-NPC | Baseline to month 18
Number of participants allocated to subprotocol AZA-001-301-GMx | Baseline to month 18

CONTACTS AND LOCATIONS:
Locations (34):
- United States (5):
  - UCSF Children's Hospital and Research Center at Oakland, Oakland, California
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Mayo Clinic Childrens Center - PIN, Rochester, Minnesota
  - Children's Medical Center Dallas, Dallas, Texas
  - Lysosomal Rare Disorders Research and Treatment Center, Fairfax, Virginia
- Argentina (2):
  - Hospital Universitario Austral, Ciudad Autónoma Buenos Aires, Buenos Aires
  - Hospital de Niños de La Santisima Trinidad, Córdoba, Córdoba Province
- Australia (3):
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Children's Hospital Melbourne - PIN, Parkville, Victoria
- Brazil (3):
  - Instituto Fernandes Figueira, Rio de Janeiro, Rio de Janeiro
  - Hospital de Clinicas de Porto Alegre (HCPA) - PPDS, Porto Alegre, Rio Grande do Sul
  - Hospital Pequeno Príncipe, Curitiba
- Canada (3):
  - M.A.G.I.C. Clinic Ltd. Metabolics and Genetics in Calgary, Calgary, Alberta
  - University of Alberta Medical Genetics Clinic, Edmonton, Alberta
  - Centre Hospitalier de l'Universite de Montreal-1000 rue Saint-Denis, Montreal, Quebec
- AP-HP - Hôpital Armand Trousseau, Paris, France
- SphinCS GmbH, Höchheim, Germany
- India (3):
  - Amrita Institute of Medical Sciences and Research Centre, Ernākulam, Kerala
  - All India Institute of Medical Sciences (AIIMS) - New Delhi, New Delhi, National Capital Territory of Delhi
  - JK Lone Hospital, Jaipur, Rajasthan
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy
- Portugal (2):
  - ULS de Santo António, EPE - Centro Materno Infantil Norte, Porto, Porto District
  - ULS de Santa Maria,EPE - Hospital de Santa Maria - PPDS, Lisbon
- Spain (2):
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona, Barcelona
  - Hospital Infantil Universitario Niño Jesus - PIN, Madrid, Madrid
- Sahlgrenska universitetssjukhuset Östra, Gothenburg, Västra Götaland County, Sweden
- Inselspital - Universitätsspital Bern, Bern, Canton of Bern, Switzerland
- Turkey (Türkiye) (3):
  - Balcali Hastanesi Saglik Uygulama ve Arastirma Merkezi, Adana, Adana
  - Gazi Universitesi Saglik Arastirma ve Uygulama Merkezi, Çankaya, Ankara
  - Ege Universitesi Tip Fakultesi, Bornova, İzmir
- United Kingdom (3):
  - Great Ormond Street Hospital, London, London
  - University College London Hospitals (UCLH), London, Middlesex
  - Royal Manchester Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No